CLINICAL TRIAL: NCT04377646
Title: A Study of Hydroxychloroquine and Zinc in the Prevention of COVID-19 Infection in Military Healthcare Workers (COVID-Milit)
Brief Title: A Study of Hydroxychloroquine and Zinc in the Prevention of COVID-19 Infection in Military Healthcare Workers
Acronym: COVID-Milit
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Military Hospital of Tunis (Other)
Collaborators: UR17DN02 : Autoimmune Diseases Research Unit (Unknown); Dacima Consulting (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UR17DN02-001; TN2020-NAT-INS-38 (Other: Tunisian Ministry of Health)
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Sars-CoV2; COVID19
Keywords: Prophylaxis; Zinc; Hydroxychloroquine; Health Professionals; Military
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Zinc

STUDY DESIGN:
Intervention Model Description: Double blind randomized clinical trial with 3 arms
Who Masked: Participant, Care Provider, Investigator
Masking Description: Random blind allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydroxychloroquine & Zinc (Active Comparator): Will receive:
  * Hydroxychloroquine 400 mg at day 1 and day 2, then a weekly dose of 400 mg up to 2 months.
  * Zinc 15 mg at daily dose up to 2 months
  Interventions: Drug: Hydroxychloroquine; Drug: Zinc
- Hydroxychloroquine (Active Comparator): Will receive:
  * Hydroxychloroquine 400 mg at day 1 and day 2, then a weekly dose of 400 mg up to 2 months.
  * Placebo of Zinc
  Interventions: Drug: Hydroxychloroquine; Drug: Zinc (Placebo)
- Placebo (Placebo Comparator): Will receive a double placebo (Hydroxychloroquine and Zinc) up to 2 months
  Interventions: Drug: Hydroxychloroquine (placebo); Drug: Zinc (Placebo)

INTERVENTIONS:
Drug: Hydroxychloroquine — 400 mg at day 1 and day 2, then 400 mg weekly up to 2 months
  Arms: Hydroxychloroquine; Hydroxychloroquine & Zinc
Drug: Hydroxychloroquine (placebo) — 1 pill at day 1 and day 2, then 1 pill weekly up to 2 months
  Arms: Placebo
Drug: Zinc — 15 mg per day up to 2 months
  Arms: Hydroxychloroquine & Zinc
Drug: Zinc (Placebo) — 1 pill per day up to 2 months
  Arms: Hydroxychloroquine; Placebo

SUMMARY:
A multicenter randomized clinical trial aiming to assess the efficacy of hydroxychloroquine associated to Zinc compared to hydroxychloroquine, in the prevention of Military Health Professionals Exposed to SARS CoV2 in Tunisia

DETAILED DESCRIPTION:
Detailed Description: The study is a multicenter randomized controlled double blind clinical trial, including up to 660 military health professionals working in Tunisia and exposed to SARS CoV2 at different levels (2 levels of exposure).

The trial will assess the efficacy of hydroxychloroquine associated to Zinc compared to hydrxyochloroquine. Randomization will be performed by IWRS (Interactive Web Response System) by random double blocs of 9 and 6.

Collected data are managed by the electronic data capture system (DACIMA Clinical Suite),according to the FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the EU GDPR (European General Data Protection Regulation), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation)

ELIGIBILITY:
Inclusion Criteria:

* No self-medication with chloroquine, hydroxychloroquine or antivirals
* COVID-19 negative diagnosis confirmed by "rapid test" and "PCR test" (Polymerase Chain Reaction test)
* No clinical symptoms suggestive of COVID-19
* Having given written consent for their participation in the study

Exclusion Criteria:

* Participation in other clinical trials for the treatment or prevention of SARS-COV-2 infection within 30 days before inclusion
* Hypersensitivity to any of the drugs or to any of its excipients.
* ECG showing rhythm disturbances, QT interval> 500 ms, conduction disturbances.
* Severe hepatic impairment.
* Concomitant treatments : colchicin, ergot of rye, pimozide, mizolastin, simvastatin, lomitapide, alfuzosin, dapoxetin, avanafil, ivabradin, eplerenone, dronedaron, quetiapine, ticagrelor, cisapride, astemizole, astemizol.
* Retinal pathology.
* Epilepsy.
* Myasthenia.
* Psoriasis.
* Methemoglobinemia.
* Porphyria.
* Pregnant or lactating women
* Contraindication to the study products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2020-05-04 (Estimated); Primary Completion 2020-05-24 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
SARS CoV2 infection | At 2 months of follow-up
  Frequency of confirmed SARS CoV2 infection

SECONDARY OUTCOMES:
COVID-19 symptoms description | At 2 months of follow-up
  Any COVID-19 related symptoms (cough, fever, headache, vomiting, nausea, dyspnea, diarrhea, smell disorder,conjunctivitis, dizziness)
Adverse Events | each month up to 2 months
  Any adverse event or serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Faida Ajili, MD, Study Chair — Military Hospital of Tunis; Nejla Mrabet, PhD, Study Director — Military Hospital of Tunis
Locations (1):
- Military Hospital of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No